CLINICAL TRIAL: NCT04196647
Title: Pilotstudy to Develop a Guideline for Hometitration With Doudopa for Patients With Parkinson Disease
Brief Title: Guideline for Hometitration With Duodopa for Parkinson Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Bo Biering-Soerensen, Attending, Rigshospitalet, Denmark
Other Study IDs: 15010036
Record Dates: First submitted 2019-06-04; First posted 2019-12-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; duodopa; pump; tele-medicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Home titration — Patients have their initial dosage titration of duodopa done in their own home, supported by one visit from nursing staff, and one video consultation a day

SUMMARY:
The purpose of this study is to

1. Create a guide for hometitration of Duodopa for patients with Parkinson's disease
2. Outline which patients could be considered for "hometitration"

DETAILED DESCRIPTION:
To start treatment with continuous intestinal levodopa infusion to the duodenum (Duodopa-pump) in patients with Idiopathic Parkinson Disease (IPD), it is usually required that the patient is hospitalised to test if Duodopa works for the patient and for the titration process to find the relevant dosage before operation and connection of the pump.

A hospitalisation is very costly. Experience shows, that this group of patients are often very stressed during hospitalisation because of noise, impaired sleep and unfamiliar surroundings. These conditions make fast and effective dosage titration very difficult, and experience also shows that the dosage often needs to be recalibrated once the patient is back home in familiar surroundings.

The use of TeleMedicin (TM) is on the rise in Denmark as well as other international health care systems.

These factors were the basis for the home-titration study where patients have their initial dosage titration done in their own home, supported by one visit from nursing staff, and one TM (video consultation) a day. The goal is to make the titration process more effective, reduce cost by treating the patient in their own home and making the patient more satisfied with the titration process.

ELIGIBILITY:
Inclusion criteria:

* Idiopathic Parkinson Disease (UK Parkinson's Disease Society Brain Bank criteria-UK PDSBB)
* Patient must be self-sufficient, or have access to support in own home (spouse, nursing home, home-nurse)
* Motivated and comfortable with home treatment and telemedicine (tablet provided by the clinic)

Exclusion Criteria:

* Patients not eligible for Duodopa-treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced parkinson, reffered to Duodopa treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 14 days after titration
  Satisfaction questionnaire specific for study. 10 questions with a scale from highly satisfied to not at all satisfied.

SECONDARY OUTCOMES:
Hoehn Yahr staging of Parkinson's disease | 2 month
  Scale to acces severity of symptoms of Parkinsons disease.
  1. Unilateral involvement only usually with minimal or no functional disability Unilateral involvement only 1.5 - Unilateral and axial involvement
  2. Bilateral or midline involvement without impairment of balance Bilateral involvement without impairment of balance 2.5 - Mild bilateral disease with recovery on pull test
  3. Bilateral disease: mild to moderate disability with impaired postural reflexes; physically independent Mild to moderate bilateral disease; some postural instability; physically independent
  4. Severely disabling disease; still able to walk or stand unassisted Severe disability; still able to walk or stand unassisted
  5. Confinement to bed or wheelchair unless aided Wheelchair bound or bedridden unless aided
Montreal Cognitive Assesment (MOCA) | 2 month
  Version 7.0, www.mocatest.org. Maximum points 30 (no sign of cognitive malfunction.
Parkinsons Disease Questionnaire 39 (PD-Q39) | 2 month
  39 questions for the patients to rate QoL in Parkinson's Disease.
Unified Parkinsons Disease Rating Scale III (UPDRS) | 2 month
  Scale on assesment of severity of disease induced symptoms. A total of 199 points represents the worst (total) disability.
Barthel-20 index | 2 month
  Version 30/11-2017, Maximum score 20.
Non-Motor Symptom Scale (NMSS) | 2 month
  Scale to identify non-motor symptoms within 9 domains, score fra 0 to 3, where 0 are no symptoms in that area and 3 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Biering-Sørensen, Director, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Neurologisk klinik, Rigshospitalet Glostrup, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Thomsen TH, Nielsen NS, Isenberg AL, Moller MH, Clausen JB, Schack Frederiksen IM, Olsen L, Javidi M, Vilhelmsen J, Olsen MK, Biering-Sorensen B. Home-Based Titration with Duodenal Infusion of Levodopa-Carbidopa Intestinal Gel in People with Parkinson's Disease: An Observational Feasibility Study. Parkinsons Dis. 2024 Apr 8;2024:5522824. doi: 10.1155/2024/5522824. eCollection 2024. PMID 38623494